CLINICAL TRIAL: NCT03995225
Title: Smartband/Smartphone-based Automatic Smoking Detection and Real Time Mindfulness Intervention
Brief Title: Smartband Mindfulness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000025082; 1R34AT010365-01 (NIH)
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smokers (Experimental): This study involves wearing a smartband to monitor, record and notify smokers of smoking events and deliver real-time brief mindfulness exercises by smartphone app. There is only one arm.
  Interventions: Behavioral: Smartband automatic smoking detection combined with brief mindfulness interventions

INTERVENTIONS:
Behavioral: Smartband automatic smoking detection combined with brief mindfulness interventions — Smartband/smartphone based automatic smoking monitoring, notification and real-time brief mindfulness interventions and learn to work mindfully with cravings and triggers rather than smoke using RAIN prior to smoking episodes.This is a 3 step intervention.

SUMMARY:
To determine treatment fidelity for a smartband/smartphone-based smoking monitoring, notification and brief mindfulness intervention.

DETAILED DESCRIPTION:
This study will test the feasibility of using a smartband to detect and track smoking and deliver brief smoking cessation interventions by smartphone app in real time. Smokers will wear a smartband to detect and notify them of smoking for 21 days and obtain individual smoking profiles; detected smoking will then trigger a "mindful smoking" exercise for the next 7 days leading up to their quit date at 30 days; after which another mindfulness exercise ("RAIN": recognize, accept, investigate and note cravings rather than smoke) will be delivered prior to each predicted smoking episode according to their individual smoking profile for 30 days post-quit.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Daily smokers (≥ 5 cigarettes per day)
* Daily smoker for at least 2 years
* Own an Android phone or iPhone
* Fluent in English as study content is currently only available in English
* >18 of 20 on the Action subscale of the Readiness to Change Questionnaire

Exclusion Criteria:

* E-cigarette use (some days/every day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Garrison, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Horvath M, Grutman A, O'Malley SS, Gueorguieva R, Khan N, Brewer JA, Garrison KA. Smartband-Based Automatic Smoking Detection and Real-time Mindfulness Intervention: Protocol for a Feasibility Trial. JMIR Res Protoc. 2021 Nov 16;10(11):e32521. doi: 10.2196/32521. PMID 34783663

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 155 participants completed onboarding and were considered enrolled and provided demographics data. Of these, 154 participants completed the baseline survey. Of these, 115 participants wore the smartband for at least one day. A modified intent to treat sample was analyzed for outcomes, defined as participants who completed onboarding and wore the smartband for at least one day (N=115).
Groups:
- Smokers: This study involves wearing a smartband to monitor, record and notify smokers of smoking events and deliver real-time brief mindfulness exercises including RAIN by smartphone app. There is only one arm.
  Smartband automatic smoking detection combined with brief mindfulness interventions: Smartband/smartphone based automatic smoking monitoring, notification and real-time brief mindfulness interventions
Period: Overall Study
Arm/Group | Smokers
Started (Completed Zoom onboarding) | 155 (Enrolled in the study and provided demographics data. Considered intent to treat.)
Baseline Survey Completed | 154
Smartband Worn for at Least 1 Day | 115
Confirmed/Denied Smoking on Smartband | 111 (Participants who wore the smartband for at least one day, and additionally confirmed/denied smoking events detected by the smartband, allowing measurement of correct detection of smoking events and false alarms.)
Received Mindful Smoking Exercise Triggered by Smoking | 114 (Participants had smoking events during the mindful smoking part of the study and therefore received mindful smoking exercises triggered by smartband-detected smoking. All participants who wore the smartband for at least one day (N=115) were able to receive mindful smoking triggered by the smartband, even if they never confirmed/denied smoking.)
21-day Survey Completed | 112
28-day Survey Completed | 101
Primary Smoking Outcomes Reported at End of Treatment | 96 (Participants who reported primary outcomes measuring smoking but did not complete the full end of treatment survey.)
End of Treatment Survey Completed | 95
Completed (Total number analyzed had to wear smartband for at least one day) | 115
Not Completed | 40

BASELINE CHARACTERISTICS:
Population: Demographics were reported at enrollment, prior to the baseline survey, and therefore are reported for the enrolled sample (N=155).
Arm/Group | Smokers
Number analyzed (Participants) | 155
Age, Customized [Mean (Standard Deviation); unit: years] | 46.06 (10.41)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 83
  Male | 71
  Female and Non-binary | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-hispanic White | 118
  Hispanic White | 3
  Black or African American | 6
  Asian | 5
  Other or Multiracial | 23
Region of Enrollment [Number; unit: participants]
  United States | 155
Education [Count of Participants; unit: Participants]
  Some College | 129
  GED/equivalent or high school or less education | 26

OUTCOME MEASURES:

1. Primary Outcome: Fidelity of Detecting Smoking Episodes
Description: Percent of smoking episodes detected and the rate of false alarms in the first 60 days of the study during which smokers are wearing the smartband to monitor, detect and notify them of smoking episodes.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: percentage of events
Arm/Group | Smokers
Number analyzed (Participants) | 111
percentage of events
  Average percent of smoking events correctly detected | 90.2 (17.5)
  Average percent of false alarms | 9.8 (17.5)

2. Primary Outcome: Fidelity of Delivering Mindful Smoking Exercises Triggered by Smoking
Description: Percent of mindful smoking exercises correctly triggered by detected smoking episodes and the rate of false alarms during which any detected and confirmed smoking event triggers the mindful smoking exercise.
Time Frame: 39 days
Measure: Mean (Standard Deviation); unit: percentage of events
Arm/Group | Smokers
Number analyzed (Participants) | 114
percentage of events
  percent of mindful smoking exercises correctly triggered | 95.6 (10.9)
  percent of false alarms | 9.8 (17.5)

3. Primary Outcome: Timeliness of Delivering RAIN Exercise
Description: Percent of participants and score range (very low, low, moderate, high, very high), with feasibility determined by 75% of participants rating timeliness of RAIN exercise as moderate or higher (via real-time ecological momentary assessment). Moderate or higher indicates a better (more timely) outcome.
Time Frame: 30 days
Population: participants who completed at least one RAIN exercise
Measure: Number; unit: percentage of participants
Arm/Group | Smokers
Number analyzed (Participants) | 84
percentage of participants
  Percent participants who rated timeliness as moderate, high or very high | 83.3
  Percent participants who rated timeliness as very low or low | 16.7

4. Primary Outcome: Adherence to Wearing the Smartband
Description: Percent of days spent wearing the smartband.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Smokers
Number analyzed (Participants) | 115
percentage of days | 69.6 (30.5)

5. Primary Outcome: Adherence to Answering Smartband Notifications of Smoking Events
Description: Percent of smoking notifications answered
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: percentage notifications answered
Arm/Group | Smokers
Number analyzed (Participants) | 111
percentage notifications answered | 98.2 (4)

6. Primary Outcome: Adherence to Answering Ecological Momentary Assessment Items
Description: Percentage of ecological momentary assessment (EMA) ratings (e.g., timeliness, helpfulness, craving, affect) answered when participants completed mindfulness exercises. That is, did the participant complete the EMA when they completed the mindfulness exercise. Measured separately for percentage of EMA answered when participants completed RAIN exercises, and percentage of EMA answered when participants completed mindful smoking exercises. Reported is the percentage of EMA answered out of the number of completed mindfulness exercises, separately for RAIN and mindful smoking.
Time Frame: 60 days
Measure: Number; unit: Percentage of ratings answered
Arm/Group | Smokers
Number analyzed (Participants) | 115
Percentage of ratings answered
  When completed RAIN exercises | 98.3
  When completed mindful smoking exercises | 100

7. Primary Outcome: Adherence to Completing Mindfulness Exercises
Description: Percent of mindfulness exercises (RAIN, mindful smoking) completed
Time Frame: 60 days
Population: Of the 115, 75 participants completed mindfulness exercises across treatment, 94 participants completed RAIN exercises across treatment
Measure: Mean (Standard Deviation); unit: percentage of exercises completed
Arm/Group | Smokers
Number analyzed (Participants) | 115
percentage of exercises completed
  mindful smoking exercises: number analyzed (Participants) | 75
  mindful smoking exercises | 40.3 (31)
  RAIN exercises: number analyzed (Participants) | 94
  RAIN exercises | 7.9 (13.9)

8. Primary Outcome: Acceptability of Intervention - Helpfulness of Mindfulness Exercises
Description: Percent of participants and score range (very low, low, moderate, high, very high), with feasibility determined by 75% of participants rating helpfulness as moderate or higher of participants that completed at least one mindful smoking or RAIN exercise.
Time Frame: 60 days
Population: Of the 115, 75 participants completed mindfulness exercises across treatment, 84 participants completed RAIN exercises across treatment
Measure: Number; unit: percentage of participants
Arm/Group | Smokers
Number analyzed (Participants) | 115
percentage of participants
  Completed at least one mindful smoking exercise and rated it as moderately or more helpful: number analyzed (Participants) | 75
  Completed at least one mindful smoking exercise and rated it as moderately or more helpful | 74.7
  Completed at least one RAIN exercise and rated it as moderately or more helpful: number analyzed (Participants) | 84
  Completed at least one RAIN exercise and rated it as moderately or more helpful | 76.2

9. Primary Outcome: Acceptability of Intervention - User Experiences Survey
Description: Feedback on user experiences survey (e.g., whether there were too many or not enough interventions) by theme- One survey with feasibility determined by 75% of participants rating the question as moderate or higher. Below are percentage of participants with ratings of moderate or higher for each question.
Time Frame: up to 60 days
Population: N based on number of participants that answered the question at each milestone out of the 115 that wore the smartband for at least one day.
Measure: Number; unit: percentage of participants
Arm/Group | Smokers
Number analyzed (Participants) | 115
percentage of participants
  Instructions for getting started with smartband were easy to follow at onboarding: number analyzed (Participants) | 112
  Instructions for getting started with smartband were easy to follow at onboarding | 110
  Easy to wear smartband every day at day 21: number analyzed (Participants) | 112
  Easy to wear smartband every day at day 21 | 101
  Helpful to be notified of their smoking events at day 21: number analyzed (Participants) | 112
  Helpful to be notified of their smoking events at day 21 | 99
  Liked being notified of their smoking events at day 21: number analyzed (Participants) | 112
  Liked being notified of their smoking events at day 21 | 104
  Being notified of smoking events helped participants pay attention to their smoking at day 21: number analyzed (Participants) | 112
  Being notified of smoking events helped participants pay attention to their smoking at day 21 | 101
  Mindful smoking exercise were helpful at day 28: number analyzed (Participants) | 101
  Mindful smoking exercise were helpful at day 28 | 80
  Mindful smoking exercise helped them pay attention to their smoking at day 28: number analyzed (Participants) | 101
  Mindful smoking exercise helped them pay attention to their smoking at day 28 | 93
  RAIN exercises were helpful at day 60: number analyzed (Participants) | 95
  RAIN exercises were helpful at day 60 | 71

10. Secondary Outcome: Number of Participants With Self-reported Abstinence From Smoking
Description: As a secondary aim we will also evaluate self-reported one-week point prevalence abstinence from smoking and prolonged abstinence from smoking (≤5 cigarettes since quit date)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Smokers
Number analyzed (Participants) | 96
Participants
  one week point prevalence | 14
  prolonged abstinence | 29

ADVERSE EVENTS:
Time Frame: up to 60 days
Groups:
- Smokers: This study involves wearing a smartband to monitor, record and notify smokers of smoking events and deliver real-time brief mindfulness exercises by smartphone app. There is only one arm.
  Smartband automatic smoking detection combined with brief mindfulness interventions: Smartband/smartphone based automatic smoking monitoring, notification and real-time brief mindfulness interventions
Arm/Group | Smokers
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03995225/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03995225/ICF_001.pdf